CLINICAL TRIAL: NCT03184623
Title: Time Course of Changes in Muscle Mass and Body Composition During ICU Admission
Brief Title: Muscle Mass and Body Composition
Status: Completed | Type: Observational
Sponsor: Frisius Medisch Centrum (Other)
Responsible Party: Principal Investigator, Matty Koopmans, research coordinator, Frisius Medisch Centrum
Other Study IDs: nWMO 205
Record Dates: First submitted 2017-06-09; First posted 2017-06-12 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Muscle Loss
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: muscle mass measurement — measurement of muscle mass by echocardiography

SUMMARY:
ICUacquired weakness is a common complication of critical illness, particularly in patients receiving mechanical ventilation and/or suffering from conditions leading to the systemic inflammatory response syndrome.

DETAILED DESCRIPTION:
The weakness and disability that result from these neuromuscular disorders can dominate the lont-term course and impede recovery.

In this observational study we try to measure muscle mass and body composition by echocardiography and BIVA at admission and on day 2, 5

ELIGIBILITY:
Inclusion Criteria:

* all acute admitted patients in ICU

Exclusion Criteria:

* age < 18
* stay on ICU < 48 hours
* use of corticosteroids
* neurological diseases
* acute kidney injure / nead of CVVH

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted to the ICU with an expected lenght of stay > 48 hours
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2017-09-05 (Actual); Study Completion 2017-09-05 (Actual)

PRIMARY OUTCOMES:
change in muscle mass measurements during ICU stay | baseline, day 2 and day 5
  measurement by echography

CONTACTS AND LOCATIONS:
Overall Officials: Matty Koopmans, MSc, Principal Investigator — MCL
Locations (1):
- Medical Center Leeuwarden, Leeuwarden, Netherlands

IPD SHARING:
Plan to Share IPD: No